CLINICAL TRIAL: NCT05308186
Title: Effectiveness of Sensory Stimulation on Attenuating Pain and Stress Among Patients With Disorders of Consciousness, Hospitalized in a Prolonged Respiratory Department- A Pilot Study
Brief Title: Effectiveness of Sensory Stimulation on Attenuating Pain and Stress Among Patients With Disorders of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Samson Assuta Ashdod Hospital (Unknown); Bet Hadar- Medical rehabilitation and nursing center (Unknown)
Responsible Party: Principal Investigator, Tami Bar-Shalita, Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0151-21-AAA
Record Dates: First submitted 2022-02-24; First posted 2022-04-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Disorder of Consciousness
Keywords: disorders of consciousness; pain; prolonged respiratory failure; sensory stimulation
MeSH Terms: conditions — Consciousness Disorders; Pain | interventions — Acoustic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The guardians and outcome assessor will not be made aware of the order of interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auditory stimulation (Experimental): Exposing the patient to an audio-based stimulus.
  Interventions: Behavioral: Auditory stimulation
- Auditory and tactile stimulations (Experimental): Combination of tactual and audio-based stimuli.
  Interventions: Behavioral: Auditory and tactile stimulations

INTERVENTIONS:
Behavioral: Auditory stimulation — The patient will be exposed to music that he used to enjoy (from the family's or guardian's report) through headphones. In case no report is given, nature (brook) sounds will be streamed.
  Arms: Auditory stimulation
Behavioral: Auditory and tactile stimulations — The patient will be exposed to music that he used to enjoy (from the family's or guardian's report, otherwise nature (brook) music will be streamed) through headphones combined with deep tissue massage will be given on the upper limbs.
  Arms: Auditory and tactile stimulations

SUMMARY:
The aim of the presented study is to examine the effectiveness of sensory stimulation in reducing pain and stress of patients diagnosed with Disorder of consciousness.

DETAILED DESCRIPTION:
Background: Disorder of consciousness (DOC) is a medical state in which the person's ability to be aware of himself and his surroundings is impaired due to an acquired brain injury. Neuroimaging during nociceptive stimulation in patients with DOC shows an activation in the network affiliated with the affective dimension of pain, providing evidence that patients can feel pain without behavioral signs. While patients not experiencing DOC receive medical care for reducing pain derived from daily medical procedures, patients with DOC receiving these same medical procedures do not receive such care for pain alleviation. Sensory stimulation has been found as an effective intervention for the stabilization and improvement of physiological signs, yet its' effectiveness in reducing pain in patients with DOC has not been studied.

Methods: Crossover experimental research will be conducted on one focus group without a control group, that includes recurring tests prior and after intervention. At the first stage of the research, the data will be collected twice a day, for fourteen days, once when the patient is in rest and once pre- and post-endotracheal suction. The second stage will include interventions based on two arms - auditory stimulation and a combination of auditory and tactile stimulations at the same time. Measures will be collected in days one, seven and fourteen in each arm. All measures will be applied pre- and post-endotracheal suction which will be conducted after the intervention period, as specified above, and during a patient rest period before and after intervention. Both interventions will be conducted for ten minutes each, twice daily, for fourteen days.

Population: After receiving consent to participate in the study from a guardian,15 adults aged 30-75, diagnosed with DOC, hospitalized in prolonged respiratory department will participate.

Tools: Physiological signs, behavioral pain scale, Modify Ashworth Scale, Brain Engagement Index.

Expected Results:

1. Statistical significance will be found between measurements prior to interventions (control) and after interventions, both during rest (clinical pain) and during medical procedures, in the following measures:

   1. Physiological signs (blood pressure, pulse and respiratory indices) post intervention will be lower.
   2. Degree of spasticity post intervention will be lower.
   3. Pain levels post intervention will be lower.
2. Statistical significance will be found in the levels of attention during interventions (sensory stimulations) in comparison to before the interventions (control), where the former will be higher in comparison to the latter.
3. Statistical significance will be found in the efficiency of multi-sensory stimulations in comparison to a single sensory stimulation, where the former will show lower physiological signs, spasticity, and levels of pain during rest and medical procedures.

Findings may improve the quality of life in patients with respiratory distress, diagnosed with DOC, providing additional treatment options for pain management other than medications.

ELIGIBILITY:
Inclusion Criteria:

* Stable vital and essential signs taken from a nurse report
* A score between 1-4 in Coma Near Coma scale.

Exclusion Criteria:

* Spinal cord injury
* Past neurological disorders
* Past psychiatric disorders
* Pressure ulcers
* Prolonged fever
* Cellulite in one limb or more
* Urine retention

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
Behavioral pain scale (BPS) change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arms 1 & 2 twice on days 1, 7, 14
  BPS evaluates three behavioral domains (facial expressions, movement of upper limbs, and compliance with ventilation) that are based on observation of the patient body's posture and his response to a nociceptive stimulation. Each subscale is scored from 1 (no response) to 4 (full response). Therefore, possible BPS scores range from 3 (no pain) to 12 (maximum pain).
Modify Ashworth scale (MAS) change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arms 1 & 2 twice on days 1, 7, 14
  MAS is used to measure the increase of muscle tone which is manifested by an increased resistance of joints to passive movement. The MAS measures on the following 6 level ordinal scale: 0 = no increased resistance; 1 = slightly increased resistance (catch followed by relaxation or minimal resistance at the end of the range of motion); 1+ = slightly increased resistance (catch followed by minimal resistance throughout less than half of the range of motion); 2 = clear resistance throughout most of the range of motion; 3 = strong resistance; passive movement is difficult; 4 = rigid flexion or extension.
EEG brainwave change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arms 1 & 2 twice on days 1, 7, 14
  EEG will be sampled using the Mind-Wave dry electrode system, with one frontal electrode and one reference electrode on the earlobe, at a sampling rate of 512Hz. Positioning of the electrode conforms with the goal of monitoring prefrontal activity, which may correlate with attention regardless of the site of lesion. The sampled data is transferred through a wireless connection to the computer, where the Brain Engagement Index (BEI) is processed in real-time every 10 seconds and presented by the BEI monitor.
Respiratory Rate (RR) change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arm 1 twice daily for 14 days; Change from baseline measured during arm 2 twice daily for 14 days
  The set ventilatory rate is the minimum number of breaths delivered to the patient per minute. The actual rate may be higher than the set rate if the patient is initiating spontaneous breaths. Rate is also a determinant of ventilation and is adjusted in response to the patient's CO2 (carbon dioxide) levels. RR will be collected from the patient's respiratory machine.
Tidal Volume (TV) change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arm 1 twice daily for 14 days; Change from baseline measured during arm 2 twice daily for 14 days
  Tidal volume (TV) is the volume of gas delivered to the patient with each breath. Tidal volume may also be expressed as TV. TV is only set for volume-controlled modes of ventilation and is usually 8-12cc/kg of body weight. TV will be collected from the patient's respiratory machine.
Peak Inspiratory Pressure (PIP) change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arm 1 twice daily for 14 days; Change from baseline measured during arm 2 twice daily for 14 days
  Inspiratory pressure reflects global alveolar pressure and is monitored continuously. The maximum allowable PIP is set on the ventilator. If the PIP exceeds the set value, an alarm will sound, and gas delivery will halt until the next breath is triggered. The normal peak inspiratory pressure on a mechanically ventilated patient with normal lungs is approximately 20cm H2O (water). The maximum allowable peak pressure varies from patient to patient. The pulmonologists determine the safest pressure for each patient. PIP values should be trended in volume-controlled modes to detect changes in pulmonary compliance. PIP will be collected from the patient's respiratory machine.
Systolic Blood Pressure (SBP) change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arm 1 twice daily for 14 days; Change from baseline measured during arm 2 twice daily for 14 days
  SBP will be measured using monitoring equipment located in the departments. A device from Philips Medical Systems will be used. USA Model Suresigns VS2 +. Cross-sectional values for systolic blood pressure: norm 120-129, normal-high 130-139, and hypertension ≥140. SBP will be collected using a monitoring equipment located in the departments.
Diastolic Blood Pressure (DBP) change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arm 1 twice daily for 14 days; Change from baseline measured during arm 2 twice daily for 14 days
  DBP will be measured using monitoring equipment located in the departments. A device from Philips Medical Systems will be used. USA Model Suresigns VS2 +. Optimal diastolic blood pressure values <80, with cross-sectional points to norm 80-84, normal-high 85-89, and hypertension ≥90. DBP will be collected using a monitoring equipment located in the departments.
Heart Rate (HR) change | Baseline is measured pre-intervention twice daily for 14 days. Change from baseline measured during arm 1 twice daily for 14 days; Change from baseline measured during arm 2 twice daily for 14 days
  HR will be measured using monitoring equipment located in the departments. A device from Philips Medical Systems will be used. USA Model Suresigns VS2 +. The average pulse value is 60-80 beats per minute. HR will be collected using a monitoring equipment located in the departments.

OTHER OUTCOMES:
Screening tool Coma Near Coma (CNC) scale | This tool will be used once as a filter to participate in research one day prior to measuring the baseline
  The CNC is a scale for patients with acquired brain injury, who function at very low levels of consciousness. The scale evaluates the occurrence of responses to visual, auditory, command following, threat response, olfactory, tactile, pain and vocalization. The CNC is both a quantitative assessment-with scores ranging from 4 (lowest level of consciousness) to 0 (highest level of consciousness)-and a qualitative assessment-with 5 levels comprising extreme coma (3.5-4), marked coma (2.9-3.49), moderate coma (2.01-2.89), near coma (0.9-2), no coma (0-0.89). Patients will be considered for the research between level 4-extreme coma to level 1-near coma.

CONTACTS AND LOCATIONS:
Overall Officials: Shely Farag Harpak, B.O.T, Study Chair — Tel Aviv University; Yoseph Mishal, Dr., Principal Investigator — Bet Hadar- Medical rehabilitation and nursing center
Locations (1):
- Bet Hadar- Medical rehabilitation and nursing center, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be available upon personal request

REFERENCES:
- See also: Validation of a behavioral pain scale in critically ill, sedated, and mechanically ventilated patients. — http://doi.org/10.1213/01.ANE.0000182331.68722.FF
- See also: Pain measurement techniques: Spotlight on mechanically ventilated patients. — https://doi.org/10.2147/JPR.S151169
- See also: Comparison of Single and Combined Effects of Nature Sounds and Foot Sole Reflexology Massage on the Level of Consciousness in Traumatic Comatose Patients — http://doi.org/10.1097/HNP.0000000000000326
- See also: Suctioning: A review of current research recommendations — http://doi.org/10.1016/S0964-3397(02)00004-6
- See also: The effects of massage and music on pain, anxiety and relaxation in burn patients: Randomized controlled clinical trial — http://doi.org/10.1016/j.burns.2017.01.011
- See also: The effect of sensory stimulation provided by family on arterial blood oxygen saturation in critical care patients — http://www.ncbi.nlm.nih.gov/pubmed/25709692
- See also: Inter-and intra-rater reliability of the Modified Ashworth Scale: A systematic review and meta-analysis — http://doi.org/10.23736/S1973-9087.17.04796-7
- See also: Assessing pain in critically ill sedated patients by using a behavioral pain scale — http://doi.org/10.1097/00003246-200112000-00004
- See also: Plum and Posner's Diagnosis of Stupor and Coma — https://books.google.co.il/books?hl=iw&lr=&id=AggSDAAAQBAJ&oi=fnd&pg=PR9&dq=Plum+and+Posner%E2%80%99s++diagnosis+of+stupor+and+coma&ots=Cq6tSgV5qV&sig=ETNN-3ALG2eMjP1L_LHmIon9Cg0&redir_esc=y#v=onepage&q=Plum%20and%20Posner%E2%80%99s%20%20diagnosis%20of%20stupor%20and%20coma&f=false
- See also: Use of Music and Voice Stimulus on Patients With Disorders of Consciousness — http://doi.org/10.1097/JNN.0b013e3182029778
- See also: Accuracy of Critical Care Pain Observation Tool and Behavioral Pain Scale to assess pain in critically ill conscious and unconscious patients: Prospective, observational study — http://doi.org/10.1186/s40560-016-0192-x
- See also: Effects of the Sensory Stimulation Program on Recovery in Unconscious Patients With Traumatic Brain Injury — http://doi.org/10.1097/JNN.0b013e3181a23e94
- See also: EEG and autonomic responses to nociceptive stimulation in disorders of consciousness — http://doi.org/10.1016/J.JOCN.2018.09.020
- See also: Psychometric Properties of the Coma Near-Coma Scale for Adults in Disordered States of Consciousness: A Rasch Analysis — http://doi.org/10.1016/j.apmr.2020.10.119